CLINICAL TRIAL: NCT07032090
Title: The Effect of Health Education Based Laughter Yoga Applied to Adolescents on Stress and Digital Gaming Habits
Acronym: Digital Habits
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, PhD, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/98
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Digital Technology; Technology Addiction; Internet Addiction Disorder; Laughter Yoga
Keywords: Laughter Yoga; Digital Technology; Technology Addiction; Internet Addiction Disorder; Adolescent; Stress; Health Education
MeSH Terms: conditions — Technology Addiction; Internet Addiction Disorder; Health Education | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: A four-arm randomized controlled study using the Solomon design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1:Health Education and Laughter Yoga (Experimental): Participants will complete a pre-test, receive a single face-to-face session of stress management education, followed by laughter yoga twice a week for 6 weeks.
  Interventions: Behavioral: Health education; Behavioral: Laughter Yoga
- Arm 3: Health Education and Laughter Yoga (Experimental): Participants will receive a single face-to-face session of stress management education without a pre-test, followed by laughter yoga twice a week for 6 weeks.
  Interventions: Behavioral: Health education; Behavioral: Laughter Yoga
- Arm 2: Control Group (No Intervention): Participants will undergo a pre-test with no additional intervention; post-tests will be conducted at the end of the study, and laughter yoga will be offered to volunteers.
- Arm 4: Control Group (No Intervention): Participants will not undergo a pre-test and no additional intervention will be provided; post-tests will be conducted at the end of the study, and laughter yoga will be offered to volunteers.

INTERVENTIONS:
Behavioral: Health education — Participants will receive face-to-face health education, followed by 12 sessions of laughter yoga.
  Other Names: stress coping training
  Arms: Arm 1:Health Education and Laughter Yoga; Arm 3: Health Education and Laughter Yoga
Behavioral: Laughter Yoga — The intervention groups will receive a total of 12 sessions of laughter yoga, delivered by the researcher over 6 weeks, twice a week, each lasting 40-45 minutes.
  Arms: Arm 1:Health Education and Laughter Yoga; Arm 3: Health Education and Laughter Yoga

SUMMARY:
Adolescents may turn to digital games as a coping mechanism for stress, which can lead to addiction and various health problems. School-based health education and laughter yoga are promising interventions for reducing stress and promoting healthy behaviors. This randomized controlled trial with a Solomon four-group design aims to evaluate the effects of health education and laughter yoga on stress levels and digital game habits among adolescents.

Study Hypotheses:

H0-1: Health education and laughter yoga have no effect on adolescent stress. H1-1: Health education and laughter yoga reduce adolescent stress. H0-2: Health education and laughter yoga do not affect digital game habits. H1-2: Health education and laughter yoga reduce digital game habits.

DETAILED DESCRIPTION:
This study is designed as a four-arm randomized controlled trial using the Solomon design. It aims to evaluate the effects of health education and laughter yoga on adolescents' stress levels and digital gaming habits. The intervention will be conducted during April-May 2025 with middle school students enrolled in grades 5 through 8.

The study sample will include 68 volunteer students who meet the inclusion criteria and provide parental consent. Participants will be assigned to four groups using stratified simple randomization: Intervention I, Intervention II, Control I, and Control II.

* Intervention I Group: Participants will complete a pre-test, receive a single-session health education on stress and coping, followed by laughter yoga sessions conducted twice weekly for six weeks (total of 12 sessions). A post-test will be administered at the end.
* Intervention II Group: Participants will receive the same health education and laughter yoga intervention without a pre-test. Post-test will be conducted after the sessions.
* Control I Group: Participants will complete the pre-test but will not receive any intervention during the study. A post-test will be applied at the end of the study, followed by an optional laughter yoga session.
* Control II Group: Participants will not complete a pre-test or receive any intervention. A post-test will be administered at the end of the study, followed by an optional laughter yoga session.

The assessment tools include the "Digital Game Addiction Scale for Children" and the "Adolescent Stress Questionnaire - Short Form." At the end of the intervention, participant satisfaction will also be assessed using group-specific satisfaction questionnaires.

Data analysis will involve descriptive statistics (frequency, percentage, mean, standard deviation) and appropriate inferential tests based on the distribution of the data. Parametric or non-parametric tests will be used as applicable. Linear models will assess the main effects of group and time, as well as the interaction between them. The significance level will be set at p<0.05.

This research is expected to contribute to school-based public health interventions by evaluating a combined strategy involving health education and a non-pharmacological stress management technique (laughter yoga) among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who are students in the 5th, 6th, 7th, and 8th grades,
* whose parents and themselves volunteer to participate in the study,
* who play digital games using devices such as mobile phones, tablets, computers, or game consoles will be included in the study.

Exclusion Criteria:

* Adolescents who have any health condition that prevents them from exercising; -who have undergone abdominal surgery within the last three months; or
* who have diabetes, glaucoma, hypertension, epilepsy, asthma,
* hernia will be excluded from the study.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Digital Game Addiction Scale for Children | 1.5 months
  It was developed by Hazar and Hazar (2017) to determine the levels of digital game addiction in children aged 10-14. The scale, prepared as a 5-point Likert type, consists of 4 sub-factors and 24 items. Each item on the scale is coded as "1 = Strongly Disagree," "2 = Disagree," "3 = Neutral," "4 = Agree," and "5 = Strongly Agree." The lowest possible score on the scale is 24, and the highest is 120. The scoring classification is as follows: "1-24: Normal group, 25-48: Low-risk group, 49-72: Risk group, 73-96: Addicted group, 97-120: Highly addicted group." The sub-dimensions of the scale are: "Excessive Focus and Conflict Related to Digital Gaming," "Tolerance Development in Game Time and Value Assigned to the Game," "Postponement of Individual and Social Tasks/Homework," and "Psychological-Physiological Reflection of Withdrawal and Immersion in the Game." The Cronbach's alpha for the entire scale is 0.90, and for the sub-factors, it is 0.78, 0.81, 0.76, and 0.67, respectively.
Adolescent Stress Questionnaire -Short Form | 1.5 month
  The Adolescent Stress Questionnaire was developed by Byrne et al. in 2007 as a 5-point Likert-type scale consisting of 58 items and 10 subscales. In 2018, Anniko et al. created a shortened version of the questionnaire with 27 items and 9 subscales. The Turkish validity and reliability study of the scale was conducted by Öztürk Tanış and Gür in 2022.
  The questionnaire asks participants to evaluate the degree to which each item represents a source of stress for them. Each item is rated on a scale from:
  "1 = Not at all stressful (or did not occur)," "2 = A little stressful," "3 = Moderately stressful," "4 = Quite stressful," "5 = Very stressful."
  Higher scores indicate higher levels of perceived stress. The Cronbach's alpha for the original version of the scale is 0.93. For the Turkish version, the overall Cronbach's alpha is 0.88, and the subscale alphas range from 0.62 to 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No